CLINICAL TRIAL: NCT05410054
Title: The Prognostic Analysis of Upper Limb Motor Dysfunction After Stroke Based on Dynamic Connection of Motion Network
Brief Title: Quantitative Prognostic Analysis of Upper Limb Motor Dysfunction After Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Ran Li, Attending physician, Fu Xing Hospital, Capital Medical University
Other Study IDs: 2022FXHEC-KY002
Record Dates: First submitted 2022-03-23; First posted 2022-06-08 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Rehabilitation; Tobacco Use; Upper Extremity Dysfunction; Prognosis; Functional MRI
MeSH Terms: conditions — Stroke; Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good prognosis: Patients with higher Fugl-Meyer motor function scale (upper limb part) and higher Action Research Arm Test (ARAT) score.
  Interventions: Other: no intervention
- poor prognosis: Patients with lower Fugl-Meyer motor function scale (upper limb part) and lower Action Research Arm Test (ARAT) score.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — observational research

SUMMARY:
30% - 66% of stroke survivors have upper limb dysfunction. Effective rehabilitation can improve the prognosis, but the rehabilitation resources are limited. How to evaluate the prognosis early and formulate an individualized rehabilitation plan based on realistic expectations is still inconclusive. The current research shows that some brain network changes are related to the recovery of motor function. The dynamic connection of multi-modal and spatio-temporal fusion of motor network is helpful to the prognosis analysis of upper limb dyskinesia after stroke. 178 stroke patients will be included in this project. Fugl-Meyer motor function scale (upper limb part) and Action Research Arm Test (ARAT) will be evaluated at enrollment, 1month/3month/6month after onset. According to the results, the groups with good prognosis and poor prognosis will be distinguished; blood oxygen level dependent imaging and diffusion tensor imaging will be collected at the same time to compare the similarities and differences of the function and structural connection of the motion network; the correlation between interhemispheric connection, intrahemispheric connection, cross network connection of motor network and prognosis will be analyzed, the clinical and imaging features of different prognosis will be extracted. This study can provide scientific data support for the prognosis analysis of upper limb dysfunction after stroke, the improvement of rehabilitation clinical decision-making and the optimization of rehabilitation resource allocation.

ELIGIBILITY:
Inclusion Criteria:

* First stroke with upper limb motor dysfunction, Stable condition; 18 ≤age≤80 years old; The onset time was less than 3 weeks at the time of enrollment; Sign informed consent.

Exclusion Criteria:

* Stroke patients with intracranial infection, multi-system atrophy and other central nervous system diseases; Combined with severe aphasia, visual spatial neglect and other cognitive impairment; Untreated spasm (Ashworth ≥ grade 2); Obvious joint contracture restricting the movement of upper limb; In vivo metal implants; Claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients with upper limb motor dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2022-08-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Motor assessment at early subacute phase | 1 month after onset
  Fugl-Meyer Assessment for Upper Limb
Motor assessment at subacute phase | 3 months after onset
  Fugl-Meyer Assessment for Upper Limb
Motor assessment at chronic phase | 6 months after onset
  Fugl-Meyer Assessment for Upper Limb
Functional assessment at early subacute phase | 1 month after onset
  Action Research Arm Test
Functional assessment at subacute phase | 3 months after onset
  Action Research Arm Test
Functional assessment at chronic phase | 6 months after onset
  Action Research Arm Test
The motion network of early subacute phase with functional MRI | 1 month after onset
  The structural and functional connection of the motion network
The motion network of subacute phase with functional MRI | 3 months after onset
  The structural and functional connection of the motion network
The motion network of chronic phase with functional MRI | 6 months after onset
  The structural and functional connection of the motion network
Correlation analysis between changes of motor function and changes of motor network | 1 month after onset, 3 months after onset, 6 months after onset
  The correlation between interhemispheric connection, intrahemispheric connection, cross network connection of motor network and motor function prognosis will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Lirong Huo, Study Director — Fu Xing Hospital, Capital Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lundquist CB, Nielsen JF, Arguissain FG, Brunner IC. Accuracy of the Upper Limb Prediction Algorithm PREP2 Applied 2 Weeks Poststroke: A Prospective Longitudinal Study. Neurorehabil Neural Repair. 2021 Jan;35(1):68-78. doi: 10.1177/1545968320971763. Epub 2020 Nov 20. PMID 33218284
- [Background] Stinear CM, Byblow WD, Ackerley SJ, Smith MC, Borges VM, Barber PA. Proportional Motor Recovery After Stroke: Implications for Trial Design. Stroke. 2017 Mar;48(3):795-798. doi: 10.1161/STROKEAHA.116.016020. Epub 2017 Jan 31. PMID 28143920
- [Background] Stinear CM. Prediction of motor recovery after stroke: advances in biomarkers. Lancet Neurol. 2017 Oct;16(10):826-836. doi: 10.1016/S1474-4422(17)30283-1. Epub 2017 Sep 12. PMID 28920888
- [Background] Hoonhorst MHJ, Nijland RHM, van den Berg PJS, Emmelot CH, Kollen BJ, Kwakkel G. Does Transcranial Magnetic Stimulation Have an Added Value to Clinical Assessment in Predicting Upper-Limb Function Very Early After Severe Stroke? Neurorehabil Neural Repair. 2018 Aug;32(8):682-690. doi: 10.1177/1545968318785044. Epub 2018 Jul 4. PMID 29972088
- [Background] Binder E, Leimbach M, Pool EM, Volz LJ, Eickhoff SB, Fink GR, Grefkes C. Cortical reorganization after motor stroke: A pilot study on differences between the upper and lower limbs. Hum Brain Mapp. 2021 Mar;42(4):1013-1033. doi: 10.1002/hbm.25275. Epub 2020 Nov 9. PMID 33165996
- [Background] Nazarova M, Kulikova S, Piradov MA, Limonova AS, Dobrynina LA, Konovalov RN, Novikov PA, Sehm B, Villringer A, Saltykova A, Nikulin VV. Multimodal Assessment of the Motor System in Patients With Chronic Ischemic Stroke. Stroke. 2021 Jan;52(1):241-249. doi: 10.1161/STROKEAHA.119.028832. Epub 2020 Dec 15. PMID 33317414
- [Background] Puig J, Blasco G, Alberich-Bayarri A, Schlaug G, Deco G, Biarnes C, Navas-Marti M, Rivero M, Gich J, Figueras J, Torres C, Daunis-I-Estadella P, Oramas-Requejo CL, Serena J, Stinear CM, Kuceyeski A, Soriano-Mas C, Thomalla G, Essig M, Figley CR, Menon B, Demchuk A, Nael K, Wintermark M, Liebeskind DS, Pedraza S. Resting-State Functional Connectivity Magnetic Resonance Imaging and Outcome After Acute Stroke. Stroke. 2018 Oct;49(10):2353-2360. doi: 10.1161/STROKEAHA.118.021319. PMID 30355087
- [Background] Lee J, Lee A, Kim H, Shin M, Yun SM, Jung Y, Chang WH, Kim YH. Different Brain Connectivity between Responders and Nonresponders to Dual-Mode Noninvasive Brain Stimulation over Bilateral Primary Motor Cortices in Stroke Patients. Neural Plast. 2019 Apr 7;2019:3826495. doi: 10.1155/2019/3826495. eCollection 2019. PMID 31093270
- [Background] Xia Y, Huang G, Quan X, Qin Q, Li H, Xu C, Liang Z. Dynamic Structural and Functional Reorganizations Following Motor Stroke. Med Sci Monit. 2021 Mar 11;27:e929092. doi: 10.12659/MSM.929092. PMID 33707406
- [Background] Simpson LA, Hayward KS, McPeake M, Field TS, Eng JJ. Challenges of Estimating Accurate Prevalence of Arm Weakness Early After Stroke. Neurorehabil Neural Repair. 2021 Oct;35(10):871-879. doi: 10.1177/15459683211028240. Epub 2021 Jul 28. PMID 34319189
- [Background] Backhaus W, Braass H, Higgen FL, Gerloff C, Schulz R. Early parietofrontal network upregulation relates to future persistent deficits after severe stroke-a prospective cohort study. Brain Commun. 2021 May 4;3(2):fcab097. doi: 10.1093/braincomms/fcab097. eCollection 2021. PMID 34056601